CLINICAL TRIAL: NCT02321748
Title: A Single-centre, Open-label, Randomised, Crossover, Drug-drug Interaction Study in Healthy Men to Investigate the Effect of a Single Dose of ASP2151 on the Pharmacokinetics of Montelukast
Brief Title: Drug-Drug Interaction Study: ASP2151 and Montelukast
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maruho Europe Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: M522101-EU23
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Results first posted 2019-01-14 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Healthy
Keywords: HSV; Herpes; volunteers; drug-drug interaction
MeSH Terms: conditions — Herpes Simplex | interventions — montelukast; ASP2151

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Montelukast (Other): 10mg montelukast alone followed by 10mg montelukast + 400mg ASP2151
  Interventions: Drug: Montelukast; Drug: ASP2151
- ASP2151 (Other): 10mg montelukast + 400mg ASP2151 followed by 10mg montelukast alone
  Interventions: Drug: Montelukast; Drug: ASP2151

INTERVENTIONS:
Drug: Montelukast
  Other Names: SINGULAIR
Drug: ASP2151

SUMMARY:
CYP2C8 is involved in the metabolism of many drugs. So, it is important to assess in vivo the inhibitory effect of ASP2151 on that enzyme to determine any possible drug interactions. The aim of this trial is to investigate the potential for interaction of ASP2151 with the CYP2C8 probe substrate montelukast.

ELIGIBILITY:
Inclusion Criteria:

* A body mass index (Quetelet index) in the range 18.0-30.9.
* Sufficient intelligence to understand the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of, the entire trial.
* Willingness to give written consent to participate after reading the information and consent form, and after having the opportunity to discuss the trial with the investigator or his delegate.
* Willingness to give written consent to have data entered into The Overvolunteering Prevention System.

Exclusion Criteria:

* Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the pre-trial screening assessment that could interfere with the objectives of the trial or the safety of the volunteer.
* Any of the following liver function tests higher than 1.5 times the ULN at the screening visit: aspartate aminotransferase (AST), alanine aminotransferase (ALT), ALP, bilirubin, gamma glutamyl transpeptidase (gamma-GT).
* Platelet counts outside normal limits.
* Presence of acute or chronic illness or history of chronic illness sufficient to invalidate the volunteer's participation in the trial or make it unnecessarily hazardous.
* Clinically significant impaired endocrine, thyroid, hepatic, respiratory or renal function, diabetes mellitus, coronary heart disease, or history of any psychotic mental illness.
* History of bleeding diathesis.
* Surgery (eg stomach bypass) or medical condition that might affect absorption of medicines.
* Presence or history of severe adverse reaction to any drug, history of multiple drug allergies (multiple defined as >3), or sensitivity to trial medication.
* Use, during the 28 days before the first dose of trial medication, of any prescription medicine, or any other medicine or herbal remedy (such as St John's wort) known to interfere with the CYP3A4, CYP2C19, CYP2C8 or CYP2C9 metabolic pathway (unless judged as not clinical significant by the investigator and sponsor). See Appendix 1: for common CYP3A4, CYP2C19, CYP2C8 and CYP2C9 interactors/substrates.
* Use, during the 7 days before the first dose of trial medication, of any over the counter medicine, with the exception of paracetamol (acetaminophen).
* Participation in another clinical trial of a new chemical entity or a prescription medicine within the previous 3 months.
* Presence or history of drug or alcohol abuse, or intake of more than 21 units of alcohol weekly or more than 10 cigarettes daily.
* Blood pressure and heart rate in seated position at the screening examination outside the ranges 90-140 mm Hg systolic, 40-90 mm Hg diastolic; heart rate 40_100 beats/min. However, if the investigator deems the result to be not clinically significant the subject may be included.
* Possibility that the volunteer will not cooperate with the requirements of the protocol.
* Evidence of drug abuse on urine testing.
* Positive test for hepatitis B, hepatitis C, HIV1 or HIV2.
* Loss of more than 400 mL blood during the 3 months before the trial, eg as a blood donor.
* Objection by General Practitioner (GP) to volunteer entering trial.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research Ltd, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at one investigative site in United Kingdom from 03-December 2014 to 01-April 2015
Groups:
- Montelukast, Then Montelukast + ASP2151: 10mg montelukast alone followed by 10mg montelukast + 400mg ASP2151
  Montelukast
  ASP2151
- Montelukast + ASP2151, Then Montelukast: 10mg montelukast + 400mg ASP2151 followed by 10mg montelukast alone
  Montelukast
  ASP2151
Period: Overall Study
Arm/Group | Montelukast, Then Montelukast + ASP2151 | Montelukast + ASP2151, Then Montelukast
Started | 12 | 12
First Intervention (4 Days) | 12 | 12
Wasout (2weeks) | 12 | 12
Second Intervention (4 Days) | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Montelukast, Then Montelukast + ASP2151 | Montelukast + ASP2151, Then Montelukast | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: year] | 28.5 (7.7) | 33.2 (5.8) | 30.8 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 12 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 9 | 10 | 19
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Concentration (Cmax) of Montelukast
Time Frame: Blood samples were taken at pre-dose of Day 1 and 0.5, 1,1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24, 30, 36, 48 and 72h after post doses in first or second intervention
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Montelukast: 10mg montelukast alone followed by 10mg montelukast + 400mg ASP2151
  Montelukast
  ASP2151
- ASP2151: 10mg montelukast + 400mg ASP2151 followed by 10mg montelukast alone
  Montelukast
  ASP2151
Arm/Group | Montelukast | ASP2151
Number analyzed (Participants) | 24 | 24
ng/mL | 415.6 (24.9) | 505.9 (25.7)

2. Primary Outcome: Time of Peak Concentration (Tmax) of Montelukast
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Montelukast | ASP2151
Number analyzed (Participants) | 24 | 24
h | 3 [2.00 to 6.00] | 3 [1.50 to 5.00]

3. Primary Outcome: Area Under the Curve (AUC) of Montelukast
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Montelukast | ASP2151
Number analyzed (Participants) | 24 | 24
h*ng/mL | 2799.2 (29.7) | 3418.5 (30)

4. Primary Outcome: Half-Life (t1/2) of Montelukast
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Montelukast | ASP2151
Number analyzed (Participants) | 24 | 24
h | 4.87 (27.8) | 5.37 (18.5)

5. Primary Outcome: Apparent Volume of Distribution (Vd/f) of Montelukast
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Montelukast | ASP2151
Number analyzed (Participants) | 24 | 24
L | 26.72 (10.482) | 23.76 (7.854)

6. Primary Outcome: Apparent Total Body Clearance (CL/f) of Montelukast
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Montelukast | ASP2151
Number analyzed (Participants) | 24 | 24
L/h | 3.72 (1.079) | 3.04 (0.857)

7. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Refer to the result of adverse event.
Time Frame: Up to 32 days after the last dose
Measure: Number; unit: participants
Groups:
- Montelukast Alone: Participants received montelukast 10 mg alone in first or second intervation
- Montelukast With ASP2151: Participants received montelukast 10 mg with ASP2151 400mg in first or second intervation
Arm/Group | Montelukast Alone | Montelukast With ASP2151
Number analyzed (Participants) | 24 | 24
participants
  Non-serious adverse event | 7 | 2
  serious adverse event | 0 | 0

8. Other Pre Specified Outcome: Peak Plasma Concentration (Cmax) of Methyl Hydroxymontelukast
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Montelukast | ASP2151
Number analyzed (Participants) | 24 | 24
ng/mL | 19.18 (40.5) | 23.28 (51.9)

9. Other Pre Specified Outcome: Time of Peak Concentration (Tmax) of Methyl Hydroxymontelukast
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Montelukast | ASP2151
Number analyzed (Participants) | 24 | 24
h | 4.51 [3.00 to 6.00] | 5 [2.50 to 6.00]

10. Other Pre Specified Outcome: Area Under the Curve (AUC) of Methyl Hydroxymontelukast
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Montelukast | ASP2151
Number analyzed (Participants) | 24 | 24
h*ng/mL | 150.19 (46.6) | 188.62 (59)

11. Other Pre Specified Outcome: Half-Life (t1/2) of Methyl Hydroxymontelukast
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Montelukast | ASP2151
Number analyzed (Participants) | 24 | 24
h | 4.87 (24.7) | 4.83 (25.3)

12. Other Pre Specified Outcome: Peak Plasma Concentration (Cmax) of ASP2151
Time Frame: Blood samples were taken at pre-dose of Day 1 and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16 and 24h after post doses in first or second intervention
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ASP2151
Number analyzed (Participants) | 24
ng/mL | 1679.7 (32.4)

13. Other Pre Specified Outcome: Time of Peak Concentration (Tmax) of ASP2151
Time Frame: as for outcome 12
Measure: Median (Full Range); unit: h
Arm/Group | ASP2151
Number analyzed (Participants) | 24
h | 3 [1.50 to 4.00]

14. Other Pre Specified Outcome: Area Under the Curve (AUC) of ASP2151
Time Frame: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | ASP2151
Number analyzed (Participants) | 24
h*ng/mL | 20928.2 (29.4)

15. Other Pre Specified Outcome: Half-Life (t1/2) of ASP2151
Time Frame: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | ASP2151
Number analyzed (Participants) | 24
h | 8.406 (17.4)

16. Other Pre Specified Outcome: Apparent Volume of Distribution (Vd/f) of ASP2151
Time Frame: as for outcome 12
Measure: Mean (Standard Deviation); unit: L
Arm/Group | ASP2151
Number analyzed (Participants) | 24
L | 246.9 (104.44)

17. Other Pre Specified Outcome: Apparent Total Body Clearance (CL/f) of ASP2151
Time Frame: as for outcome 12
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | ASP2151
Number analyzed (Participants) | 24
L/h | 19.95 (6.525)

ADVERSE EVENTS:
Time Frame: Up to 32 days after the last dose
Groups:
- Montelukast: Participants received montelukast 10 mg alone in first or second intervention
- ASP2151: Participants received montelukast 10 mg with ASP2151 400mg in first or second intervention
Arm/Group | Montelukast | ASP2151
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 7/24 | 2/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Montelukast (N=24) | ASP2151 (N=24)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Gingivitis (Infections and infestations) | 1 | 0
Nasopharynｇitis (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No